CLINICAL TRIAL: NCT05046730
Title: SEAM Trial: Sutureless End to End Anastomosis by Magnetic Compression: A Study to Evaluate Safety and Effectiveness of Self-Forming Magnet (SFM) Anastomosis Device: A Historically Controlled Propensity Matched Study
Brief Title: SEAM Trial: Sutureless End to End Anastomosis by Magnetic Compression
Acronym: SEAM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruiting
Sponsor: GI Windows, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: GIW 21-002
Record Dates: First submitted 2021-09-08; First posted 2021-09-16 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Retraction of Ileostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Prospective Evaluation of the SFM Device (Experimental): This is a multicenter, single-arm study in which clinical outcomes prospectively evaluated for a minimum of 100 subjects undergoing ileostomy reversal using the SFM Anastomosis Device
  Interventions: Device: Ileostomy Reversal using Self Forming Magnets (SFM)
- Retrospective Chart Review of Historical Controls (Active Comparator): In order to have a sufficient pool of retrospective patients for matching, retrospective data will be collected for a minimum of 300 patients. The historical control cohort will be accrued from the same pool of institutions participating in the prospective study.
  Interventions: Device: Ileostomy Reversal using Self Forming Magnets (SFM)

INTERVENTIONS:
Device: Ileostomy Reversal using Self Forming Magnets (SFM) — The magnets will be manually deployed into the small intestine during open surgery following creation of a mini or full laparotomy as clinically indicated. Once the desired segment of small bowel is resected, the magnet is inserted through the open ends of each bowel section. Once proper magnet position is confirmed and the bowel ends are approximated, the magnets couple to form the anastomosis.

SUMMARY:
The objectives of this study are to determine the safety and effectiveness of the SFM Anastomosis Device when used to create a small bowel anastomosis for patients undergoing ileostomy reversal as compared with a propensity-matched historic control group of patients who underwent ileostomy reversal using a conventional closure technique (sutures or stapler).

DETAILED DESCRIPTION:
This is a multicenter, single-arm study in which clinical outcomes prospectively evaluated for a minimum of 100 subjects undergoing ileostomy reversal using the SFM Anastomosis Device will be 1:1 propensity score matched through nearest neighbor matching to a historical control cohort of patients who underwent ileostomy reversal using conventional closure techniques. In order to have a sufficient pool of retrospective patients for matching, retrospective data will be collected for a minimum of 300 patients. The historical control cohort will be accrued from the same pool of institutions participating in the prospective study. Eligibility criteria will be standardized between the prospective investigational treatment arm and the historical control. Within this analysis, propensity score (PS) matching will be used to reduce bias due to potential differences in key covariates between the prospective and retrospective cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be >18 years
2. Participant has a temporary loop ileostomy that was created ≥ 2 months but ≤ 10 months prior to reversal. NOTE: The inclusion of patients with ileostomy after total colectomy and palliative ileostomy is permitted if the patients have estimated overall survival of greater than 2 years or if the loop ileostomy is resulting in persistent fluid and electrolyte disorders or other significant stoma related complications where closure of the ileostomy is required for patient safety.
3. Preoperative clearance with confirmation of anastomotic integrity of the original resection; i.e., absence of active exacerbation of inflammatory disease (as applicable), stricture or leakage at or distal to the diverted colorectal anastomosis via gastrografin enema and/or endoscopy based on physician's discretion
4. BMI ≤ 40 kg/m2
5. American Society of Anesthesiologist (ASA) score < IV at time of reversal
6. All cancer patients must have completed chemotherapy ≥2 months prior to ileostomy closure
7. Subject or authorized representative have been informed of the nature of the study and has provided written informed consent approved by the appropriate local Institutional Review Board (IRB) and agrees to comply with all protocol-specified follow-up appointments

Exclusion Criteria:

1. Radiological or clinical signs of anastomosis leak, active infection (except uncomplicated urinary tract infection)
2. Ongoing or prolonged ileus or bowel obstruction from original surgery
3. Requires/d additional abdominal surgery (e.g., Major hernia repair, either necessitating mesh and/or abdominal wall reconstruction) after ileostomy or requires/d concurrent abdominal surgery during reversal procedure
4. Multiple small bowel obstructions occurring between ileostomy creation and closure requiring a formal abdominal exploration through a midline incision at the time of ileostomy closure or any other participant in whom laparotomy is required at time of ileostomy closure
5. Requires/d laparotomy at time of ileostomy closure
6. Congestive heart failure with ejection fraction<35% or clinically significant arrhythmia (any rhythm disturbances except sinus tachycardia, sinus bradycardia or a sinus rhythm with premature atrial or ventricular complexes)
7. Decompensated chronic obstructive lung disease
8. Pulmonary embolism or myocardial infarction in the prior 6 months
9. Congenital or acquired anomalies of the gastrointestinal tract, including atresias, stenosis, luminal distortion or malrotation
10. Coagulation deficiency not normalized by medical treatment or platelet count <50,000/µL at time of reversal
11. Known moderate to severe renal disease (eGFR < 44 milliliters per minute per 1.73m2) or ongoing dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Achieving anastomosis success | 30 days
  The primary effectiveness hypothesis is that anastomosis success rate for the SFM device will be non-inferior to the anastomosis success rate observed for the propensity-matched historical control group

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Messaris, MD, Ph.D, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (14):
- United States (14):
  - Advent Health, Orlando, Florida
  - Colon and Rectal Clinical of Orlando, Orlando, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Spectrum Health / Ferguson Clinic, Grand Rapids, Michigan
  - Trinity Health Michigan Heart, Ypsilanti, Michigan
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - The Mount Sinai Medical Center, New York, New York
  - St Francis Hospital, Roslyn, New York
  - Novant Health Clinical Research, Winston-Salem, North Carolina
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Health Science Center at Houston, Houston, Texas
  - The Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No
No: There is not a plan to make IPD available.